CLINICAL TRIAL: NCT03395496
Title: Comparison of Biodentine and MTA Pulpotomies in the Primary Molar Teeth 3 Year Follow up
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mine Koruyucu, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-24692
Record Dates: First submitted 2017-12-26; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Pulpotomy; Dental Caries
Keywords: pulpotomy; pediatric dentistry; primary molars
MeSH Terms: conditions — Dental Caries | interventions — tricalcium silicate; TheraCal

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biodentine (Experimental): Dental materials
  Interventions: Drug: Biodentine; Drug: ProRoot (Aggregate)
- ProRoot MTA (Experimental): Dental Materials
  Interventions: Drug: Biodentine; Drug: ProRoot (Aggregate)

INTERVENTIONS:
Drug: Biodentine — Biodentine pulpotomy agent
  Other Names: 77509635
Drug: ProRoot (Aggregate) — ProRoot MTA pulpotomy agent
  Other Names: 75896452

SUMMARY:
The aim of this study is to compare two pulpotomy medicaments in primary molars clinically.A total of 200 primary molars with deep caries were treated with two different pulpotomy medicaments (Mineral Trioxide Aggregate and BiodentineTM) in this study. The inclusion criteria for tooth selection were no clinical and radiographic evidence of pulp pathology. During 36 months of follow-up at 3-month intervals, clinical and radiographic success and failures were recorded.

ELIGIBILITY:
Inclusion Criteria:

* no clinical and radiographic evidence of pulp pathology,
* no clinical and radiographic symptoms,
* no history of spontaneous pain and tenderness,
* no percussion, swelling or sinus tracts and pathologic mobility.

Exclusion Criteria:

* any clinical or radiographic evidence of pulp degeneration (spontaneous or nocturnal tooth pain, tenderness to percussion, pathological mobility, internal or external root resorption, swelling or fistula, widened periodontal ligament (PDL)
* furcal or periapical radiolucency teeth requiring more than 5 minutes to achieve hemostasis during clinical procedure.
* without permanent successor

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Total success rate | 12 months after pulpotomy treatment

SECONDARY OUTCOMES:
Total success rate | 24 months after pulpotomy treatment

OTHER OUTCOMES:
Total success rate | 36 months after pulpotomy treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided